CLINICAL TRIAL: NCT01966640
Title: Basophil Activation Test (BAT) Sensitivity in Child Food Allergy
Acronym: TAB-TPO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012/170/HP
Record Dates: First submitted 2013-10-11; First posted 2013-10-21 (Estimated); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Allergy to Egg; Allergy to Peanut
Keywords: diagnosis of allergy; Basophil Activation Test
MeSH Terms: conditions — Peanut Hypersensitivity | interventions — Basophil Degranulation Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Child food allergy suspicion (Experimental): Basophil Activation Test realized in case of Child food egg and peanut allergy suspicion
  Interventions: Biological: Basophil Activation Test

INTERVENTIONS:
Biological: Basophil Activation Test — blood sample for Basophil Activation Test

SUMMARY:
Child food allergy represent 6 to 8% of child in industrialised country. Within this allergy, peanuts and egg allergy are one of the most common.

Actually when there is a suspicion of food allergy, the OPT is the gold standard for the diagnosis. During the OPT we give increasing doses of the allergen to the patient and evaluate threshold causing a clinical reaction. This test is associated with a risk of strong allergic reaction and need a medical supervision.

Standard allergy test, like skin test or specific IgE test, can't be use for the diagnosis of these allergy. Some publications demonstrate that these tests lack sensibility and specificity for child food allergy diagnosis.

New tests have to be develop to diagnosis child food allergy without risks. The BAT is a cellular test able to evaluate the basophiles activation by specific allergen in vitro. This test allow us to evaluate more physiologically the sensitization of patients to an allergen. It is already used in drug allergy and it has been evaluated in infant milk allergy in an other clinical trial.

In this study we want to evaluate the sensitivity of BAT to the diagnosis of child food allergy compare to the gold standard test OPT. We will evaluate the BAT on 140 children with food allergy and compare this results with the OPT at the same time. If the BAT results can predict the sensitivity of children to food allergen, it could limit the use of the OPT and reduce the risk of this test.

DETAILED DESCRIPTION:
Child food allergy represent 6 to 8% of child in industrialised country. One third of these child will develop severe reactions and one third will experience multiple allergy. In France, there is few epidemiologic data but in 2005 F. Rancé evaluated the prevalence of these allergy to 6.7% of school child. Within the food allergen, peanut, egg and milk are the most common.

Currently, there is two diagnostic possibilities:

* A strong allergic reaction with identified allergens and specific IgE positive, making it highly probable diagnosis.
* A moderate allergic reaction with only suspicion on the allergen, without definitive diagnosis.

When there is a suspected allergy, the gold standard to the diagnosis is the OPT. This test consist of the gradual ingestion of the suspected food allergen to evaluate the threshold causing a clinical reaction. The OPT must be performed under medical supervision in a hospital due to the risk of severe allergic reaction.

The OPT is the gold standard in allergy diagnosis. The other tests (prick test, IgE specific measure…) are not sensitive enough. Furthermore, the level of IgE specific was not related to the risk to develop clinical reaction to the food allergen. Some studies have try to combine skin tests with the result of IgE specific measure but the sensitivity did not improve enough.

New tests have to be develop to diagnosis child food allergy without risks. The BAT is a cellular test able to evaluate, in blood, the basophiles activation by specific allergen in vitro. This test measure by flow cytométrie the expression of activation molecule (CD63) on basophiles (CCR3+) after incubation with the allergen. If the patient is sensitize to the allergen, the percentage of active basophiles will be higher than in non sensitize people. This test allow us to evaluate more physiologically the sensitization of patients to an allergen. This test has already been tested for drug allergy and milk allergy in child. This clinical trial demonstrated that in mill allergy, the BAT had a good sensitivity (91% and sensibility (96%). Furthermore, this study could determined the threshold of the BAT in child food allergy (6% of activated basophiles).

In light of these results, we want to evaluate the advantage of BAT compare to OPT in child with allergy to egg or peanut.

During this study, we will perform BAT on a blood sample from child suspected of food allergy (egg or peanut) before OPT and we will compare its results with the OPT results. The primary objective of this study is to evaluate the BAT interest to predict the results of OPT by analysing the sensibility, specificity, positive predictive value, negative predictive value of BAT.

If these study demonstrate that BAT can predict OPT results for child food allergy, we will be able to reduce the number of OPT for these patients and reduce the risk of anaphylactic shock during OPT.

ELIGIBILITY:
Inclusion Criteria:

* Child older than 6 months and less than 18 years old
* Diagnosis of type I allergy to peanut or egg
* oral provocation test to peanut or egg programmed

Exclusion Criteria:

* No possibility to assess blood sample

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Actual)
Dates: Start 2013-09-12 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2019-01-11 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the Basophil Activation Test | Day 1
  Sensitivity of the BAT compare to OPT with a threshold value of 6% for the BAT in a population of child food allergy.
  Sensitivity is defined as the capacity for BAT to have a positive result when OAT result is also positive (diagnosis of allergy confirmed)

SECONDARY OUTCOMES:
Evaluation of the proportion of child positive to the BAT | Day 1
  Evaluation of the proportion of child positive to the BAT within child positive to the OPT in the group egg allergy Evaluation of the proportion of child positive to the BAT within child positive to the OPT in the group peanut allergy

CONTACTS AND LOCATIONS:
Overall Officials: Laure COUDERC, Dr, Principal Investigator — UH Rouen
Locations (1):
- UH Rouen, Rouen, France